CLINICAL TRIAL: NCT04071041
Title: Effect of Albumin Administration on Outcomes in Hypoalbuminemic Patients Hospitalized With Community-acquired Pneumonia (ALBUCAP): a Prospective, Randomized, Phase III Clinical Controlled Trial.
Brief Title: Effect of Albumin Administration in Hypoalbuminemic Hospitalized Patients With Community-acquired Pneumonia.
Acronym: ALBUCAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Jordi Carratala (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Sponsor-Investigator, Jordi Carratala, Sponsor, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-INF-ALBUCAP-402; 2018-003117-18 (EudraCT Number); PI17/01332 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2019-07-31; First posted 2019-08-28 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Community-acquired Pneumonia; Hypoalbuminemia
Keywords: Community-acquired Pneumonia; Albumin; Inflammation
MeSH Terms: conditions — Community-Acquired Pneumonia; Hypoalbuminemia; Inflammation | interventions — Serum Albumin, Human; Albumins

STUDY DESIGN:
Intervention Model Description: A superiority, non-blinded, multicentre, randomized, interventional controlled clinical trial. Patients will be randomly assigned (1:1) to receive standard of care plus albumin (20g in 100ml) every 12 hours for 4 days or standard of care alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care plus albumin (Experimental): Patients will receive human albumin 20%, 20g in 100ml (Albutein Instituto Grifols, S.A. Can Guasch 2, Parets del Vallès, 08015 Barcelona, Spain) intravenously every 12 hours for 4 days or until death, discharge or clinical stability if occurring before.
  Patients will receive empirical antibiotic therapy according to guidelines as soon as CAP is confirmed. All microbiological assessments and additional treatment (e.g. oxygen, bronchodilators, corticosteroids, analgesic drugs, vasoactive agents, fluid resuscitation, and mechanical ventilation) will be at the discretion of the treating physicians (not the study investigators). The time of discharge and duration of antibiotics will not be determined by the study investigators, but by the treating physician team.
  Interventions: Drug: Albumin Human
- Standard care alone (No Intervention): Patients will receive empirical antibiotic therapy according to guidelines as soon as CAP is confirmed. All microbiological assessments and additional treatment (e.g. oxygen, bronchodilators, corticosteroids, analgesic drugs, vasoactive agents, fluid resuscitation, and mechanical ventilation) will be at the discretion of the treating physicians (not the study investigators). The time of discharge and duration of antibiotics will not be determined by the study investigators, but by the treating physician team.

INTERVENTIONS:
Drug: Albumin Human — Administration of albumin 20%, 20g in 100ml (Albutein Instituto Grifols, S.A. Can Guasch 2, Parets del Vallès, 08015 Barcelona, Spain) intravenously every 12 hours for 4 days or until death, discharge or clinical stability if occurring before.
  Other Names: Albutein
  Arms: Standard care plus albumin

SUMMARY:
Community-acquired pneumonia (CAP) remains a leading cause of death world-wide. Hypoalbuminemia is associated with worse outcomes. However, whether albumin administration would have a beneficial effect in outcome in patients with CAP remains uncertain.

This project proposes to test the hypothesis of whether the administration of albumin in hypoalbuminemic patients with CAP would increase the proportion of clinical stable patients at day 5.

DETAILED DESCRIPTION:
This project will consist of a superiority, non-blinded, multicentre, randomized, phase 3, interventional controlled clinical trial. The estimated sample size is of 360 patients, who will be recruited from three Spanish hospitals. Hypoalbuminemic (≤30g/L) adult patients with CAP will be randomly assigned (1:1) to receive standard care plus albumin (20g in 100ml) every 12 hours for 4 days or standard care alone.

The primary endpoint will be the proportion of clinical stable patients at day 5, defined as stable vital signs for at least 24h, analyzed by intention to treat.

The secondary endpoints will be time to clinical stability; duration of intravenous and total antibiotic treatment; length of hospital stay; intensive care unit admission; duration of mechanical ventilation and vasopressor treatment; adverse events; readmission within 30 days and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of CAP (Chest radiography consistent with CAP AND the presence of ≥2 following prespecified clinical criteria: Fever or hypothermia; Cough; Purulent sputum; High white blood cell count; Dyspnea; Pleuritic chest pain; Signs consistent with pneumonia on chest auscultation)
* Serum albumin concentration ≤ 30 g/L at presentation

Exclusion Criteria:

* Pregnancy or lactation
* Immunosuppression (e.g. chemotherapy or radiotherapy within 90 days, immunosuppressive drugs, corticosteroids at a minimum dose of 15mg/day of prednisone within 2 weeks of enrolment, HIV with a CD4 count below 200, solid organ transplant recipients, hematopoietic cell transplant recipients).
* Severe clinical status with expected survival of less than 24h.
* Congestive heart failure (New York Heart Association classes 3 or 4)
* Any contraindication for albumin administration such as hypersensitivity to albumin.
* Clinical conditions in which there is another indication for albumin administration (e.g. hepatic cirrhosis with ascites, malabsorption syndrome and nephrotic syndrome).
* Absence or impossibility of obtaining informed consent from the patient/next of kin.
* Patient already included in another clinical trial testing a treatment method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
The proportion of clinical stable patients at day 5, measured from hospital admission. | Day 5±1 of hospitalization
  Clinical stability will be defined as achieving normal oral intake, normal mental status (or usual level of functioning) and stable vital signs for at least 24 h, as previously described by Halm et al 1998

SECONDARY OUTCOMES:
Time to clinical stability (days) measured from hospital admission | Up to 30 ±5 days after discharge
  The time (days) to clinical stability, measured from hospital admission
Duration of intravenous and total antibiotic treatment (days). | Up to 30 ±5 days after discharge
  The duration of intravenous and total duration of antibiotic treatment (measured in days)
Length of hospital stay (days). | Up to hospital discharge - a median of 10 days
  The total length of hospital stay (measured in days)
Proportion of patients with intensive care unit (ICU) admission. | Up to hospital discharge - a median of 10 days
  The number of patients admitted to intensive care. For those admitted to ICU we will record: time to discharge from ICU; duration of vasopressor treatment; duration of mechanical ventilation
The rate of nosocomial infection during hospitalization | Up to hospital discharge - a median of 10 days
  The proportion of patients with nosocomial infection during hospitalization will be registered, the type of nosocomial infection will be described
Proportion of adverse events. | Up to 30 ±5 days after discharge
  Any adverse event, its severity and its possible relationship to the study drug will be assessed
The number of patients with hospital readmission within 30 days of discharge | Up to 30 ±5 days after discharge
  We will document hospital readmission within 30 days of discharge
All-cause mortality | Up to 30 ±5 days after discharge
  5-day mortality, 30-day mortality and mortality within 30 days of hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rombauts, Principal Investigator — Institut d'Investigació Biomèdica de Bellvitge; Jordi Carratalà, Study Director — Hospital Universtari de Bellvitge, Universitat de Barcelona
Locations (3):
- Spain (3):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Residència Sant Camil, Sant Pere de Ribes, Barcelona
  - SCIAS-Hospital de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rombauts A, Abelenda-Alonso G, Simonetti AF, Verdejo G, Meije Y, Ortega L, Clemente M, Niubo J, Ruiz Y, Gudiol C, Tebe C, Videla S, Carratala J. Effect of albumin administration on outcomes in hypoalbuminemic patients hospitalized with community-acquired pneumonia (ALBUCAP): a prospective, randomized, phase III clinical controlled trial-a trial protocol. Trials. 2020 Aug 20;21(1):727. doi: 10.1186/s13063-020-04627-1. PMID 32819439